CLINICAL TRIAL: NCT05870202
Title: Optimizing Diabetes Care Quality for Low-Income Patients
Brief Title: Treatment Burden Screening Questionnaire Pilot Study
Acronym: TBQ
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: Hennepin Health Care (Unknown)
Responsible Party: Sponsor
Other Study IDs: GIM-2024-33207
Record Dates: First submitted 2023-04-28; First posted 2023-05-23 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Type 2 Diabetes
Keywords: type 2 diabetes; treatment burden
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Potentially Inappropriate Medication List

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: screening tool — The screening tool identifies areas of treatment burden in patients with type 2 diabetes. The tool is in the form of a brief questionnaire that the patient completes prior to a clinical appointment. The patient's responses to the questionnaire are then included in the discussion with the patient's primary care clinician during the clinical visit.

SUMMARY:
The main objective of this study is to develop and evaluate a clinic-based pilot intervention to optimize patient-centered diabetes care for low income patients at risk for low quality diabetes care and poor outcomes.

DETAILED DESCRIPTION:
Single arm trial of a brief screening tool to identify areas of treatment burden in patients with diabetes, which will then be used as a tool in a primary care clinician visit discussion. We will assess (primary outcome) the acceptability and feasibility of 1. recruitment and retention processes; 2. screening tool usability; and (secondary outcomes) 3. outcome assessments. Data will include systematic tracking of recruitment and retention efforts, baseline and follow-up participant data, post-visit surveys of clinicians and participants, and patient participant qualitative interviews.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older, a diagnosis of T2DM, receiving primary care in a participating clinic, and having an in-person clinic visit with a participating trained clinician.

Exclusion Criteria:

* Cognitive impairment, residing in a nursing home, and pregnancy (to avoid recruiting patients with gestational diabetes).

Ages: 18 Years to 95 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients with type 2 diabetes receiving care in a safety-net primary care clinic.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2023-03-07 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of the clinical trial | Baseline to 6 month follow up
  Patients' willingness to participate in the study as assessed by:
  1) percentage of approached and eligible patients who consent to enroll in the study, 2) percentage of participants who completed the study procedures including baseline survey data collection, 3) use of the screening tool and completion of the post-intervention visit survey 4) time (days) to recruit 50 subjects across 2 clinic sites.
Acceptability | Baseline to 6 month follow up
  Helpfulness and utility of the intervention screening tool as assessed by 1) patient post intervention surveys and clinician post intervention surveys to identify patterns of patient and clinician participants' impressions of the helpfulness and utility of the intervention, and 2) acceptability of the intervention using qualitative interviews.

SECONDARY OUTCOMES:
Change in HbA1c | Baseline and 6 month follow up
  Change in HbA1c from baseline to 6 months

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Community University Health Center, Minneapolis, Minnesota
  - Hennepin Health Care - Whittier Clinic, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: No